CLINICAL TRIAL: NCT05693181
Title: Systemic Administration of Allogenic Mononuclear Cord Blood Cells in Patients With Acute Severe Contusion Spinal Cord Injury: Safety and Efficiency Evaluation, Stages I/II
Brief Title: Cord Blood Cells in Patients With Acute SCI
Acronym: SUBSCI II
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Collaborators: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other); K.L. Hetagurov North-Osetian State University (Unknown)
Responsible Party: Principal Investigator, Vladimir A. Smirnov, Senior researcher, M.D., Ph.D., Sklifosovsky Institute of Emergency Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 007-2022
Record Dates: First submitted 2022-11-21; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injury, Acute
Keywords: spinal cord injury; SCI; neurological deficit; stem cells; cell therapy; regenerative; paraplegia; tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Neurologic Manifestations; Paraplegia; Quadriplegia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the experimental group will obtain 4 systemic (i.v.) infusions of allogenic group- and rhesus-compatible non-related mononuclear cord blood cell samples (500 +/- 50 x 10'6 cells each).
  Participants in the control group will obtain the similar volume of vehicle (sterile saline).
  Participant's devision will be performed in a randomized manner. Randomization will be performed using standard randomization computer table.
  All participants will be blinded concerning the therapy mode.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cell Therapy (Experimental): Patients having acute severe contusion spinal cord injury (cervical, thoracic or upper-lumbar) and ASIA A/B neurological deficit, within 7 days post-SCI, after primary decompressive and stabilizing surgery. All participants meet inclusion and exclusion criteria. All participants obtain 4 infusions of allogenic non-related group- and rhesus-compatible mononuclear cord blood cells samples (500 +/- 50 x 10*6 cells each) with a 1-week interval. All participants are followed up for 12 months post-SCI.
  Interventions: Biological: Multiple systemic (i.v.) administration of allogenic non-related group- and rhesus-compatible mononuclear cord blood cells
- Vehicle (Placebo Comparator): Patients having acute severe contusion spinal cord injury (cervical, thoracic or upper-lumbar) and ASIA A/B neurological deficit, within 7 days post-SCI, after primary decompressive and stabilizing surgery. All participants meet inclusion and exclusion criteria. All participants obtain 4 infusions of vehicle (sterile saline) with a 1-week interval. All participants are followed up for 12 months post-SCI.
  Interventions: Other: Control vehicle (sterile saline)

INTERVENTIONS:
Biological: Multiple systemic (i.v.) administration of allogenic non-related group- and rhesus-compatible mononuclear cord blood cells — Each HUCBCs sample contain 500 +/- 50 x 10*6 allogenic non-related group- and rhesus-compatible mononuclear cord blood cells
  Arms: Cell Therapy
Other: Control vehicle (sterile saline) — Sterile saline infusion in control patients
  Arms: Vehicle

SUMMARY:
This is a prospective, single-blinded, single-center, randomized, comparative, interventional clinical study of systemic mononuclear multiple allogenic cord blood cells administration safety and efficiency in patients having acute severe contusion spinal cord injury (ASIA A/B), phase I/II

DETAILED DESCRIPTION:
Phase I/II of the SUBSCI II (Systemic Umbilical Cord Blood Administration in Patients with Acute Severe Contusion Spinal Cord Injury II) study is focused on safety and primary efficacy of multiple systemic infusions of allogeneic unrelated human umbilical cord blood mononuclear cells in patients with severe acute spinal cord contusion having severe neurologic deficit (ASIA A/B).

In a previous clinical study (SUBSCI I/IIa) complete safety and significant efficiency of systemic administration of human umbilical cord blood cells (HUCBCs) was demonstrated. Current study is established to confirm and verify the obtained results in a larger group of patients.

SUBSCI II study includes 80 patients with acute severe contusion spinal cord injury (SCI) and American Spinal Injury Association (ASIA) level A/B deficit divided into 2 groups (experimental and control groups, 40 patients in each). Patients will be treated with 4 infusions of group-matched and rhesus-matched cord blood samples following primary decompressive and stabilizing surgery within 7 days after SCI. All patients will be followed up for 12 months after SCI.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females, 18 to 75 years old
* Contusion spinal cord injury (SCI) at cervical, thoracic or upper lumbar (cone level) levels
* admission by 7 days post-SCI
* spinal cord contusion confirmed using MRI (T1- and T2-weighted images, STIR)
* ASIA A/B neurological deficit
* identical level of neurological deficit at admission and at the moment of patient inclusion
* primary decompressive and stabilizing surgery performed within 5 days post-SCI and prior to the first cell sample infused
* patient is ready to participate and fulfill the requirements of the study protocol
* informed consent signed by the patient or his legal representative

Exclusion Criteria:

* motor function preserved in lower limbs at admission (LEMS > 0 points) corresponding to ASIA C, D or E deficit level
* any spinal cord injury different from contusion (tear, defibering, concussion, SCIWORA, SCIWONA) confirmed using MRI
* severe combined trauma (ISS > 35 points)
* inability to perform primary decompressive and stabilizing surgery within 5 days post-SCI and prior to the first cell sample infused
* persistent systolic arterial pressure (AP) > 185 mmHg or diastolic AP > 105 mmHg or need of aggressive AP lowering using systemic antihypertensive medication at the moment of patient inclusion
* acute myocardial infarction
* blood glucose level < 3.5 Mmol/L or >21 Mmol/L or ineffective antidiabetic therapy for 24 hours
* acute or deterioration of chronic diseases of central nervous system (CNS) (e.g. stroke, non-traumatic subarachnoid hemorrhages and others at the discretion of investigator)
* hypotension or cardiovascular shock AND systolic AP < 90 mmHg OR need for intensive systemic inotropic therapy at the moment of patient inclusion
* objective need for artificial ling ventilation (ALV) at admission or prior to the stage I surgery
* acute kidney failure or deterioration of chronic kidney failure (creatinin level > 250 mumol/L or carbamide level > 25 Mmol/L)
* liver failure (general bilirubin level > 25 mumol/L, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels > 4 times exceeding upper reference limit)
* other significant disorders of vital functions
* acute of deterioration of chronic diseases of internal organs preventing from cell samples infusion
* autoimmune diseases (active or anamnestic) preventing from cell samples infusion
* allergic reactions of any type for any component of HUCBC samples
* pregnancy or lactation
* significant surgeries or severe traumas within 3 months prior to patient inclusion
* acute or chronic infection diseases (tuberculosis, lues, HIV, hepatitis B, hepatitis C etc.)
* moderate or severe hematological and/or oncohematological diseases preventing from the cell samples infusion
* any malignant tumors (both operated and not operated) or benign tumors (not operated or not totally removed) at the moment of patient inclusion
* neurological and/or psychiatric diseases preventing patient from complete understanding of study protocol or fulfillment of the study protocol requirements
* other reasons preventing patient from complete understanding of study protocol or fulfillment of the study protocol requirements
* patient's participation in any other clinical trials or studies within 6 months prior to inclusion
* immunosuppressive therapy obtained by the patient for any reason at admission
* allergic reaction for full blood or blood component transfusion in the past
* need for extracorporal detoxication methods application (hemodialysis, plasmapheresis, sorption etc.)
* bone marrow or internal organs (both donor and relative) transplantation in the past
* patient's participation in any studies applying regenerative technologies (grow factors, cytokines, cell therapy, gene therapy etc.) within 1 year prior to inclusion
* patient's rejection to sign the informed consent
* any other reasons preventing patient's inclusion according to the investigator's opinion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Continuously for 12 months post-SCI
  All adverse events (AEs) are registered within follow-up period. All registered AEs are classified using CTCAE classification and relation to the performed therapy.
Motor function | Change from Baseline 12 months post-SCI
  Evaluation of motor function dynamics in upper (UEMS), lower (LEMS) and all (GEMS) limbs
Neurological deficit | Change from Baseline 12 months post-SCI
  Evaluation of general neurological deficit dynamics using ASIA scale

SECONDARY OUTCOMES:
Sensory function | Change from Baseline 12 months post-SCI
  Evaluation of pain, tactile, temperature and proprioceptive sensory function dynamics below SCI level and comparison between two groups
Neuropathic pain syndrome | 12 months post-SCI
  Evaluation of neuropathic pain syndrome dynamics and comparison between two groups
Independent verticalization and motion ability | Change from Baseline 12 months post-SCI
  Evaluation of Independent verticalization and motion ability dynamics and comparison between two groups
Limb muscle spasticity | Change from Baseline 12 months post-SCI
  Evaluation of limb muscle spasticity level dynamics using modified Ashworth or Tardieu scales and comparison between two groups
Psychological status | Change from Baseline 12 months post-SCI
  Evaluation of psychological status dynamics using Beck depression and anxiety scales and comparison between two groups
Pelvic functions | Change from Baseline 12 months post-SCI
  Evaluation of pelvic functions dynamics (bladder fulfillment feeling, independent urination ability, urodynamic examination)
Life quality | Change from Baseline 12 months post-SCI
  Evaluation of life quality level in two groups using FIM (Functional Independence Measurement) scale and SF36 questionnaire
Electrophysiology parameters | 12 months post-SCI
  Assessment of electrophysiology objective parameters (electroneuromyography parameters with transcranial magnetic stimulation - full block, partial block or no block; somatosensory evoked potentials, motor evoked potentials)
Cell immunization | 12 months post-SCI
  Assessment of patient's immunization to infused cell samples

CONTACTS AND LOCATIONS:
Locations (1):
- N.V. Sklifosovsky Emergency Care Institute, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Personal contacts via E-mail or phone after the completion of the study